CLINICAL TRIAL: NCT02121639
Title: An Open Label Phase I/Randomised, Double Blind Phase II Study in Metastatic Castration Resistant Prostate Cancer of AZD5363 In Combination With Docetaxel and Prednisolone Chemotherapy (ProCAID)
Brief Title: Open Label Phase I/Randomised,Double Blind Phase II Study in mCRPC of AZD5363 In Combination With DP Chemotherapy
Acronym: ProCAID
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Collaborators: AstraZeneca (Industry); Cancer Research UK (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RHMCAN0935
Record Dates: First submitted 2014-04-16; First posted 2014-04-23 (Estimated); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Prostate Cancer
Keywords: Metastatic Castration Resistant Prostate Cancer; AZD5363; Docetaxel; Prednisolone
MeSH Terms: conditions — Prostatic Neoplasms | interventions — capivasertib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AZD5363 (Experimental): AZD5363
  Interventions: Drug: AZD5363
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo
  Arms: Placebo
Drug: AZD5363
  Arms: AZD5363

SUMMARY:
The aim of the ProCAID study is to determine if the addition of the AKT inhibitor AZD5363 to docetaxel and prednisolone (DP) prolongs progression free survival (PFS) in Metastatic castration resistant prostate cancer to a degree worthy of further investigation

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically proven mCRPC with documented metastases (measurable or evaluable disease is acceptable) now eligible for treatment with docetaxel chemotherapy
2. Disease progression since the last change in therapy defined by one or more of the following according to the Prostate Cancer Working Group (PCWG2) criteria (J Clin Oncol 2008;26:1148-1159):

   i. PSA progression as defined by the prostate cancer working group (2) (PCWG2) criteria (Scher et al. 2008 J Clin Oncol. 26; 1148). This must be based on a series of at least 3 readings at least 7 days apart. The 3rd reading must be >= 2ng/ml. In the event where an intermediate reading is lower than a previous reading, then the patient will still be eligible (ie. the 3 readings do not need to be consecutive). The first of the three readings must have been obtained after commencing the previous systemic therapy, or, in the case of androgen receptor antagonists, after discontinuing.

   ii. Radiographic progression of nodal or visceral metastases as defined by RECIST version 1.1 (Eur J Cancer 2009;45:228). See Appendix 5 iii. The appearance of two or more new bony metastases
3. Serum testosterone <1.7 nmol/L (ongoing LHRH analogue or antagonist therapy is permitted to maintain a castrate state)
4. Discontinuation of prior therapies for prostate cancer ≥ 4 weeks prior to commencing study treatment (with the exception of an LHRH agonist or antagonist where required for ongoing testosterone suppression)
5. No current anti-androgen withdrawal response from bicalutamide or flutamide. Consistent with PCWG2 guidelines, investigators should evaluate patients to exclude withdrawal response for 6 weeks after stopping bicalutamide or flutamide. Investigators need not wait to assess for withdrawal response in patients who did not respond, or who showed a PSA decline for ≤ 3 months, after bicalutamide or flutamide was administered as a second-line or later intervention.
6. ECOG performance status 0 or 1
7. Hb ≥ 9g/dL; platelets ≥ 100 x 109/L; neutrophils ≥ 1.5 x109/L
8. Bilirubin ≤ ULN ; ALT and AST ≤ 1.5 x ULN
9. Sodium and potassium within the normal range for the site
10. Able to swallow study drugs (without crushing/opening in the case of AZD5363)
11. Life expectancy > 3 months
12. Aged 18 years or over
13. Provision of written informed consent

Exclusion Criteria:

1. Previous treatment with cytotoxic chemotherapy for castrate resistant prostate cancer. Patients may have received previous docetaxel for up to 6 cycles given in the 'hormone sensitive setting' or ongoing bisphosphonates or denosumab. There are no restrictions on prior use of second generation hormonal therapies e.g. abiraterone, enzalutamide as long as they have been discontinued ≥ 2 weeks prior to commencing study treatment.
2. Prior malignancy with an estimated ≥ 30% chance of relapse within 2 years following curative treatment
3. Previously identified brain metastases, or spinal cord compression unless treated with full functional recovery
4. Prior radiotherapy to > 30% of bone marrow
5. Administration of an investigational agent within 30 days of first dose of study medication
6. Patients will be excluded with any of:

   i. Diabetes mellitus type I ii. Fasting plasma glucose [fasting is defined as no calorific intake for at least 8 hours] of either ≥ 7.0mmol/L (126 mg/dL) for those patients without a pre-existing diagnosis of Type 2 diabetes mellitus or ≥ 9.3 mmol/L (167mg/dL) for those patients with a pre-existing diagnosis of Type 2 diabetes mellitus iii. Glycosylated haemoglobin (HbA1C) ≥8.0% (63.9 mmol/mol) iv. Requirement for insulin for routine diabetic management and control v. Requirement for more than two oral hypoglycaemic medications for routine diabetic management and control.
7. Malabsorption syndrome, previous gastrointestinal surgery, or other gastrointestinal condition that may affect drug absorption
8. Coronary artery bypass graft, angioplasty, vascular stent, myocardial infarction, angina pectoris or congestive heart failure (NYHA ≥ grade 2) within the last 6 months
9. Abnormal echocardiogram or MUGA (LVEF should be normal according to the criteria used within the treating institution
10. Uncontrolled hypotension (systolic blood pressure <90 mmHg and/or diastolic blood pressure <50 mmHg)
11. QTc interval of >480 msec at two or more time points within a 24 hour period
12. Proteinuria (either 3+ on dipstick analysis or >500 mg/24 hours) or creatinine >1.5 x ULN concurrent with creatinine clearance <50 mL/min (assessed as per local practice e.g. by Cockcroft and Gault estimation)
13. Exposure to potent inhibitors or inducers of CYP3A4 or CYP2D6 or substrates of CYP3A4 within 2 weeks before the first dose of study treatment (3 weeks for St John's Wort)
14. Unresolved toxicity ≥ grade 2 (except alopecia) from previous cancer therapy
15. Patients with a partner of child-bearing potential who are not using a highly effective method of contraception, who are unwilling to use condoms during the study and for 30 days after the last dose of study drug
16. Known hypersensitivity to AZD5363, its excipients, or drugs in its class
17. Previous exposure to agents with the following mechanisms of action:

    * inhibition of AKT (e.g., MK2206, GDC0068, GSK2110183, GSK2141795)any inhibitor with PI3K pharmacology (e.g., GDC0941, XL147, BKM120, PX866, BYL719, AMG319, GDC0032, INK1117, INK119)
    * any compound with mixed PI3K and mammalian target of rapamycin (mTOR) kinase pharmacology (e.g., BEZ235, GDC0980, PF04691502, PF05212384, GSK2126458, XL765)
    * or any mTOR kinase inhibitor (e.g., AZD8055, AZD2014, OSI027, INK128) Note: Do not exclude patients previously treated with a rapalogue (allosteric inhibitor of mTOR; mTORC1 complex inhibitor) - including temisirolimus (Torisel; Pfizer), everolimus (Affinitor; Novartis), ridoforolimus (Ariad).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2014-01-29 (Actual); Primary Completion 2020-10-08 (Actual); Study Completion 2021-09-13 (Actual)

PRIMARY OUTCOMES:
Phase I:Determination of a suitable dose of AZD5363 | Up to 18 months
  Phase I:Determination of a suitable dose of AZD5363 using a 4 days on/3 days off continuous schedule, in combination with Docetaxol and prednisolone chemotherapy
Phase II: Progression free survival | 5 years
  Phase II: Progression free survival (PFS) in patients receiving AZD5363 versus placebo when combined with Docetaxol and prednisolone chemotherapy (DP) in metastic castration resistant prostate cancer (mCRPC)

SECONDARY OUTCOMES:
Phase I: Safety and tolerability profiles | Up to 18 months
  Phase I: Safety and tolerability profiles using Common Terminology Criteria for Adverse Events (CTCAE) version 4.03
Phase I: AZD5363 pharmacokinetics Area Under Curve (AUC) Time Frame: predose, 2, 4, 8, 24,144 hours post-dose | Up to 18 months
  Phase I: AZD5363 pharmacokinetics in combination with Docetaxol and prednisolone chemotherapy
Phase II: Bone Pain | 5 years
  Phase II: Bone pain changes using the brief pain inventory
Phase II: Progression Free Survival | 5 years
  Phase II: Progression Free Survival excluding biochemical (Prostate Specific Antigen - PSA) alone progression
Phase II: Biochemical (PSA) response rates according to PCWG2 criteria | 5 years
  Phase II: Biochemical (Prostate Specific Antigen - PSA) response rates according to Prostate Cancer Working Gourp (PCWG2) criteria
Phase II: Safety and tolerability profiles using CTCAE version 4.03 | 5 years
  Phase II: Safety and tolerability profiles using Common Terminology Criteria for Adverse Events (CTCAE) version 4.03

CONTACTS AND LOCATIONS:
Locations (1):
- Southampton General Hospital, Southampton, Hampshire, United Kingdom

REFERENCES:
- [Derived] Crabb SJ, Griffiths G, Marwood E, Dunkley D, Downs N, Martin K, Light M, Northey J, Wilding S, Whitehead A, Shaw E, Birtle AJ, Bahl A, Elliott T, Westbury C, Sundar S, Robinson A, Jagdev S, Kumar S, Rooney C, Salinas-Souza C, Stephens C, Khoo V, Jones RJ. Pan-AKT Inhibitor Capivasertib With Docetaxel and Prednisolone in Metastatic Castration-Resistant Prostate Cancer: A Randomized, Placebo-Controlled Phase II Trial (ProCAID). J Clin Oncol. 2021 Jan 20;39(3):190-201. doi: 10.1200/JCO.20.01576. Epub 2020 Dec 16. PMID 33326257
- [Derived] Crabb SJ, Birtle AJ, Martin K, Downs N, Ratcliffe I, Maishman T, Ellis M, Griffiths G, Thompson S, Ksiazek L, Khoo V, Jones RJ. ProCAID: a phase I clinical trial to combine the AKT inhibitor AZD5363 with docetaxel and prednisolone chemotherapy for metastatic castration resistant prostate cancer. Invest New Drugs. 2017 Oct;35(5):599-607. doi: 10.1007/s10637-017-0433-4. Epub 2017 Feb 1. PMID 28144789